CLINICAL TRIAL: NCT04675216
Title: Posterior Fossa Intracranial Pressure (ICP) Measurement in Cases of Traumatic, Ischemic, or Tumor Pathology (Post-surgical) at This Level: Clinical Study
Brief Title: Posterior Fossa Intracranial Pressure (ICP) Measurement: Clinical Study
Acronym: Postfossa ICP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 19/07/2017
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Pressure Increase
Keywords: Intracranial pressure; Posterior fossa; Posterior fossa tumor; Cerebellar hematoma; Cerebellar infarct
MeSH Terms: conditions — Intracranial Hypertension; Infratentorial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Posterior fossa lesion: This group will be integrated by patients with posterior fossa lesion that likely to rise the posterior fossa intracranial pressure
  Interventions: Procedure: Posterior fossa intracranial pressure measurement
- Post-operative posterior fosa surgical patients: This group will be integrated by patients operated for posterior fossa lesions in which we will try to find out what range of posterior fossa pressure is to be expected in this situation
  Interventions: Procedure: Posterior fossa intracranial pressure measurement

INTERVENTIONS:
Procedure: Posterior fossa intracranial pressure measurement — Measurement of posterior fossa pressure in an invasive way

SUMMARY:
In modern medicine, doctors attempt to monitor all physiological variables to assess their evolution and to decide, based on their changes, the therapeutic attitudes to adopt. Furthermore, this helps to establish a forecast of the evolution to be expected.

The measurement of Intracranial Pressure (ICP) has become indispensable for managing brain pathology at the anterior and middle fossa level. Doctors generally carry out this measurement at the frontal level. However, experimental and clinical studies have shown that supra-tentorial ICP measurement does not precisely predict the ICP situation in the posterior fossa.

The increased ICP in the posterior fossa is directly responsible for the clinical deterioration and eventual death in patients with tumour, hemorrhagic, or ischemic pathology of the posterior fossa structures. Some of these lesions are treatable, and their effects reversible if the increase in ICP in the posterior fossa is controlled by pharmacological or even surgical means, preventing it from reaching high levels. This need for on-time ICP control is genuine in the cerebellar hemispheres' lesions, not so much in lesions involving the brainstem. Therefore, the increase in ICP in the posterior fossa needs to be known and documented to facilitate decision-making regarding the therapy to be adopted, be it medical or surgical.

It is known what the abnormal ICP levels are at the supratentorial level, but what is not known whether these same levels apply to the posterior fossa. In other words, what it is not know with certainty is whether the same levels of ICP in the posterior fossa and its elevation during the same time are going to have equally pernicious effects or these effects are greater or lesser. Doctors need to have tables of ICP values in the posterior fossa to help them decide when these values are in the physiological range. When posterior fossa intracranial pressure lye in the pathological range, and patients need pharmacological treatment or surgical decompression, knowing for sure the posterior fossa ICP is essential. Finally, when doctors also need to know when any therapeutic attempt is useless.

Currently, doctors only monitor the ICP at the supra-tentorial level and deduce the changes in the posterior fossa from the CT and MRI images, that is, the size of the lesions, the occlusion of the cisterns, the internal cerebral hernias (cerebellar tonsils, trans-tentorial hernia from bottom to top). However, doctors do not have a tool that can objectify the pathophysiological situation of the posterior fossa's structures in real-time.

Monitoring the posterior fossa ICP will help doctors in decision-making in patients with traumatic, hemorrhagic, ischemic, or tumour pathologies (in the latter case, in the postoperative period of posterior fossa tumours). This posterior fossa ICP measurement will lead to improvements in morbidity/mortality in this subgroup of patients.

DETAILED DESCRIPTION:
The purpose of our study is to register the posterior fossa pressure in normal postoperative conditions and in patients with different kinds of posterior fossa pathologies. The aim of the study is to get a range of posterior fossa intracranial pressure values in physiological situations and then to get the same data in patients with posterior fossa pathologies. The ideal would be to monitor the posterior fossa ICP in normal subjects but this is something that does not seem ethically correct. That is why, instead, the posterior fossa ICP will be measured in posterior fossa post-operative time. These patients will have to be operated any way for their posterior fossa pathologies, and adding a posterior fossa ICP sensor does not seem a problem from the ethical point of view. In any case, patients will be asked to sign informed consent. The second aim of our study will be to compare the supratentorial (frontal area) ICP monitoring with the posterior fossa ICP monitoring to see if their values coincide or if there are deviations. This will help doctors to decide when posterior fossa ICP must be done and not to rely only on supratentorial (frontal) ICP monitoring.

1. A study will be done on 12 patients. The series published to date are very short.
2. Inclusion criteria: age 18 years, traumatic pathology, tumour, ischemic or hemorrhagic posterior fossa, GCS 8 or lower.
3. EXCLUSION CRITERIA coagulation disorders, fault multi-organic, multiple pathologies, head trauma open posterior fossa with output nerve tissue.
4. Inserting PIC level sensor above-tentorial (1 sensor PIC) and another level infra-tentorial (2nd sensor PIC).
5. Verification that the ICP sensor in the posterior fossa can be implanted at the same point as we implanted it in cadavers without more significant clinical repercussions than those seen with the insertion of the ICP at the supra-tentorial level. In that sense, we have to confirm the technique's safety at the selected point away from the lateral sinus and sigmoid sinus and the lateral part of the occipital shell. We must also verify that it is not incredibly annoying for patients (in any case, it will be patients in a coma and probably sedated), but it is about confirming that the movements of the patients do not cause problems in the ICP sensor of the posterior fossa and if they do will be sought (in collaboration with the manufacturer) technical amendments necessary to avoid any problems that go detecting
6. Data Collection ICP level supra and infra-tentorial. These data will be recorded continuously on a computer for later analysis.
7. Data analysis ICP supra and infra-tentorial comparing the figures obtained in the two compartments (the supra and infra-tentorial).
8. Analysis of the correlation or non-correlation between the supra-tentorial ICP and infra-tentorial ICP figures.
9. Correlating data PIC infra-tentorial with the clinical status of patients and their evolution.
10. Analysis of possible complications attributable to the inclusion of the ICP monitor posterior fossa, analyzing possible areas for improvement to minimize any possible risk. In particular, we will analyze the risk of bruising-hematoma in the cerebellar hemisphere at the insertion point.
11. Analysis of therapeutic decisions based on figures from the PIC in the posterior fossa.
12. Analysis of the results and their correlation with therapeutic attitudes adopted.
13. Preparation of recommendations.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years
* traumatic, tumor, ischemic, or hemorrhagic pathology of the posterior fossa
* GCS of 8 or less.

Exclusion Criteria:

* coagulation disorders
* multi-organ failure
* multiple pathologies
* open head trauma to the posterior fossa with leakage of nervous tissue

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with posterior fossa lesions, traumatic, neoplastic, ischemic, or hemorrhagic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Posterior fossa intracranial pressure | 1 month
  We will measure the posterior fossa intracranial pressure inserting a ICP sensor at the frontal area and another at the posterior fossa 2cm behind and at the level of the tip of mastoid process. The ICP values will be measured while patients are in ICU and for 2 days once back in the neurosurgical ward
Clinical status of patients | 1 month
  We will correlate the clinical status of each patient with his/her posterior fossa intracranial pressure. The clinical status will include the Glasgow Coma Scale and the Glasgow Coma Score

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General Universitario de Valencia, Valencia
  - Vicente Vanaclocha, Valencia

IPD SHARING:
Plan to Share IPD: No
To collect all the data and publish them

REFERENCES:
- [Result] Mizunari T. [Clinical aspects and intracranial pressure monitoring in cases of traumatic posterior fossa hematoma]. Nihon Ika Daigaku Zasshi. 1990 Aug;57(4):334-43. doi: 10.1272/jnms1923.57.334. Japanese. PMID 2229331
- [Result] Oshorov AV, Savin IA, Goriachev AS, Popugaev KA, Lubnin AIu. [Monitoring of intracranial pressure difference between supra- and infratentorial spaces after posterior fossa tumor removal (case report)]. Anesteziol Reanimatol. 2011 Jul-Aug;(4):74-7. Russian. PMID 21957628
- [Result] Rosenwasser RH, Kleiner LI, Krzeminski JP, Buchheit WA. Intracranial pressure monitoring in the posterior fossa: a preliminary report. J Neurosurg. 1989 Oct;71(4):503-5. doi: 10.3171/jns.1989.71.4.0503. PMID 2795169
- [Result] Rieger A, Rainov NG, Sanchin L, Ebel H, Furka I, Gorombey Z, Burkert W. Is it useful to measure supratentorial ICP in the presence of a posterior fossa lesion? Absence of transtentorial pressure gradients in an animal model. Br J Neurosurg. 1999 Oct;13(5):454-8. PMID 10627774
- [Result] Rooker S, De Visscher G, Van Deuren B, Borgers M, Jorens PG, Reneman RS, van Rossem K, Verlooy J. Comparison of intracranial pressure measured in the cerebral cortex and the cerebellum of the rat. J Neurosci Methods. 2002 Sep 15;119(1):83-8. doi: 10.1016/s0165-0270(02)00183-8. PMID 12234639
- [Result] Park CK. Accuracy of ICP monitoring in posterior fossa lesions. J Neurosurg. 1990 May;72(5):832-3. No abstract available. PMID 2324809
- [Result] Slavin KV, Misra M. Infratentorial intracranial pressure monitoring in neurosurgical intensive care unit. Neurol Res. 2003 Dec;25(8):880-4. doi: 10.1179/016164103771954014. PMID 14669535
- [Result] Wolfla CE, Luerssen TG, Bowman RM, Putty TK. Brain tissue pressure gradients created by expanding frontal epidural mass lesion. J Neurosurg. 1996 Apr;84(4):642-7. doi: 10.3171/jns.1996.84.4.0642. PMID 8613857